CLINICAL TRIAL: NCT02001688
Title: Phase II, Double-Blind, Placebo-Controlled Study to Explore the ELF and Plasma Concentration as Well as Safety of Inhaled Alpha-1 Antitrypsin in Alpha-1 Antitrypsin Deficiency Subjects
Brief Title: Phase II, Safety and Efficacy Study of Kamada-alpha-1-antitrypsin (AAT) for Inhalation"
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kamada, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Kamada-AAT (inhaled)-006
Record Dates: First submitted 2013-11-24; First posted 2013-12-05 (Estimated); Results first posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2019-12

CONDITIONS: Alpha-1 Antitrypsin Deficiency
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency | interventions — Inhalation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- Kamada-AAT for Inhalation, 80mg (Experimental): Daily inhalation of Kamada-AAT for Inhalation, 80mg
  Interventions: Drug: Kamada-AAT for Inhalation, 80mg
- Placebo (Placebo Comparator): Placebo administered by inhalation daily
  Interventions: Drug: Placebo
- Kamada-AAT for Inhalation, 160mg (Experimental): Daily inhalation of Kamada-AAT for Inhalation, 160mg
  Interventions: Drug: Kamada-AAT for Inhalation, 160mg

INTERVENTIONS:
Drug: Kamada-AAT for Inhalation, 80mg
  Arms: Kamada-AAT for Inhalation, 80mg
Drug: Placebo
  Arms: Placebo
Drug: Kamada-AAT for Inhalation, 160mg
  Arms: Kamada-AAT for Inhalation, 160mg

SUMMARY:
To evaluate different doses of "Kamada-AAT for Inhalation" on the levels of alpha 1-proteinase inhibitor and other analytes in epithelial lining fluid (ELF) and serum and to assess the safety of the treatment in subjects with AAT Deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients between 18 and 65 years of age (inclusive).
* Able and willing to sign informed consent.
* Males, and non-pregnant, non-lactating females whose screening pregnancy test is negative and who are using contraceptive methods deemed reliable by the investigator or who are post-menopausal or surgically sterilized.
* Diagnosis of alpha1-antitrypsin deficiency [only individuals with a ZZ or Z null classification].
* Forced expiratory volume in one second (FEV1) ≥ 50% of predicted post bronchodilator
* No respiratory exacerbations within 6 weeks of baseline. Subjects can be re-screened if exacerbations exist at the time of enrollment.
* No signs of chronic and/or acute Hepatitis A, Hepatitis B, Hepatitis C, HIV infection and Parvovirus B19, by NAT (for Parvovirus B19, nucleic acid testing (NAT) result must be < 10^4 IU/mL).
* No significant abnormalities in serum hematology, serum chemistry, serum inflammatory / immunogenic markers and urinalysis.
* No significant abnormalities in ECG.
* Not on intravenous augmentation therapy for at least 8 weeks prior to initial dosing with study drug/placebo and willing to forego intravenous augmentation therapy for the duration of the study.

Exclusion Criteria:

* Clinically significant intercurrent illnesses (except for respiratory or liver disease secondary to AAT deficiency), including: cardiac, hepatic, renal, endocrine, neurological, hematological, neoplastic, immunological, skeletal or other) that in the opinion of the investigator, could interfere with the safety, compliance or other aspects of this study. Patients with well-controlled, chronic diseases could possibly be included after consultation with the treating physician and the sponsor.
* History of life threatening allergy, anaphylactic reaction, or systemic response to human plasma derived products.
* History of life threatening transfusion reactions.
* History of lung transplant.
* Current or previous (up to 8 weeks from baseline) use of AAT augmentation therapy or by any other route
* Current use of oral or parenteral glucocorticoids in doses exceeding 10mg of prednisone daily or equivalent generics (substance and dose).
* Any lung surgery within the past two years.
* On any thoracic surgery waiting list.
* Active smoking during the last 12 months from screening date.
* Pregnancy or lactation.
* Woman of child-bearing potential not taking adequate contraception deemed reliable by the investigator.
* Presence of psychiatric/ mental disorder or any other medical disorder which might impair the patient's ability to give informed consent or to comply with the requirements of the study protocol.
* Evidence of alcohol abuse or history of alcohol abuse or illegal and/or legally prescribed drugs.
* Immunoglobulin A (IgA) Deficiency.
* Inability to undergo bronchoscopy.
* Allergy to lidocaine or any other medicines used in the bronchoscopy process
* Exacerbation of chronic obstructive pulmonary disease (COPD) in the previous 6 weeks.
* Participation in another clinical trial involving investigational medication or interventional treatment within 30 days prior to baseline visit.
* Participation in observational clinical trial which involves any invasive procedure scheduled to occur during the AAT inhaled study period. If participating in an observational clinical trial that already completed all diagnostic procedures (e.g. liver biopsy), any adverse events (AEs) experienced must have returned to baseline within 30 days prior to baseline visit.
* Inability to attend scheduled clinic visits and/or comply with the study protocol.
* Any other factor that, in the opinion of the investigator, would prevent the patient form complying with the requirements of the protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-04; Primary Completion 2016-02 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Florida, Pulmonary, Critical Care & Sleep Medicine, Gainesville, Florida
  - The University of Texas Health Science Center at Tyler Center for Clinical Research, Tyler, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 2 clinical sites. At each site, 18 subjects were recruited and randomized 2:1 to receive either "Kamada-AAT for Inhalation" 80 mg/day (site 1) or 160 mg/day (site 2) or placebo. This gave a total of 12 patients randomized to receive 80 mg/day active drug, 12 patients randomized to receive 160 mg/day active drug, and 12 patients placebo
Pre-assignment Details: There were no pre-assignment changes
Groups:
- Placebo: Placebo inhaled daily
Period: Overall Study
Arm/Group | Kamada-AAT for Inhalation, 80mg | Kamada-AAT for Inhalation, 160mg | Placebo
Started | 12 | 12 | 12
Completed | 12 | 11 | 11
Not Completed | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: ITT population
Groups:
- Total: Total of all reporting groups
Arm/Group | Kamada-AAT for Inhalation, 80mg | Kamada-AAT for Inhalation, 160mg | Placebo | Total
Number analyzed (Participants) | 12 | 12 | 12 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (8.69) | 55.3 (10.13) | 56.3 (4.77) | 55.7 (7.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 8 | 24
  Male | 3 | 5 | 4 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White Non-Hispanic | 12 | 12 | 12 | 36
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 12 | 12
BMI [Mean (Standard Deviation); unit: kg/m^2] | 30.0 (4.3) | 28.3 (8.3) | 25.8 (4.5) | 28.0 (6.1)
%Predicted forced expiratory volume in one second (FEV1) [Mean (Standard Deviation); unit: %] | 81.7 (17.9) | 73.2 (20.1) | 78.1 (20.0) | 77.6 (19.1)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Concentration of Antigenic Alpha-1 Antitrypsin (AAT) in the Lung Epithelial Lining Fluid (ELF)
Description: Patients underwent bronchoalveolar lavage (BAL) prior to initiation of drug and then again after 3 months. Concentration of AAT in the BAL was measured by an enzyme linked immunosorbent assay (ELISA) specific for the normal form of AAT (piM). Urea was also measured in order to determine the dilution factor of the BAL fluid and calculate the concentration of AAT in the ELF.
Time Frame: 12 weeks from initiation of study drug
Population: Intention to treat (ITT) population with values available in BAL at baseline and 12 weeks
Measure: Median (95% Confidence Interval); unit: nmol
Groups:
- Placebo: Combined placebo results from patients at the two clinical sites
Arm/Group | Kamada-AAT for Inhalation, 80mg | Kamada-AAT for Inhalation, 160mg | Placebo
Number analyzed (Participants) | 12 | 10 | 10
nmol | 4551.023 [2587 to 6835.6] | 13454.772 [1020.7 to 70907.95] | -27.15 [-103.6 to 196.7]
Statistical Analysis 1: Comparison: Kamada-AAT for Inhalation, 80mg vs Placebo; Test type: Superiority; p = 0.0005, Wilcoxon (Mann-Whitney) — One-sided test was used for antigenic and functional AAT levels to maintain overall 2.5% level of significance
Statistical Analysis 2: Comparison: Kamada-AAT for Inhalation, 160mg vs Placebo; Test type: Superiority; p = 0.020, Wilcoxon (Mann-Whitney); One-sided test was used for antigenic and functional AAT levels to maintain overall 2.5% level of significance
Statistical Analysis 3: Comparison: Kamada-AAT for Inhalation, 80mg vs Kamada-AAT for Inhalation, 160mg; Test type: Superiority; p = 0.0192, Wilcoxon (Mann-Whitney); One-sided test was used for antigenic and functional AAT levels to maintain overall 2.5% level of significance

2. Primary Outcome: Change From Baseline to 12 Weeks in the Concentration of Functional AAT (Alpha-1 Antitrypsin) in ELF
Description: ITT population with baseline and 12 week values. Patients underwent bronchoalveolar lavage (BAL) prior to initiation of drug and then again after 3 months. Concentration of AAT in the BAL was measured by an antineutrophil elastase capacity (ANEC) assay. Urea was also measured in order to determine the dilution factor of the BAL fluid and calculate the concentration of AAT in the ELF.
Time Frame: 12 weeks from initiation of study drug
Measure: Median (95% Confidence Interval); unit: nmol
Arm/Group | Kamada-AAT for Inhalation, 80mg | Kamada-AAT for Inhalation, 160mg | Placebo
Number analyzed (Participants) | 12 | 10 | 10
nmol | 2766.343 [840.9 to 3800.3] | 3557.563 [1582.8 to 10673.2] | 5.831 [-1032 to 884.3]
Statistical Analysis 1: Comparison: Kamada-AAT for Inhalation, 80mg vs Placebo; Test type: Superiority; p = 0.0005, Wilcoxon (Mann-Whitney) — One-sided test was used for antigenic and functional AAT levels to maintain overall 2.5% level of significance; p-value of Stratified Wilcoxon test
Statistical Analysis 2: Comparison: Kamada-AAT for Inhalation, 160mg vs Placebo; Test type: Superiority; p = 0.0193, Wilcoxon (Mann-Whitney); One-sided test was used for antigenic and functional AAT levels to maintain overall 2.5% level of significance
Statistical Analysis 3: Comparison: Kamada-AAT for Inhalation, 80mg vs Kamada-AAT for Inhalation, 160mg; Test type: Superiority; p = 0.2485, Wilcoxon (Mann-Whitney); One-sided test was used for antigenic and functional AAT levels to maintain overall 2.5% level of significance

3. Secondary Outcome: Change From Baseline in Levels of M Specific AAT in Plasma (PiM)
Description: Intention to treat (ITT) population with baseline and 12 week values.The median change from baseline to Week 12 in the levels of M-specific AAT (piM) in plasma was measured using a specific ELISA assay for M-specific AAT (piM)
Time Frame: 12 weeks from initiation of study drug
Measure: Median (95% Confidence Interval); unit: nM
Arm/Group | Kamada-AAT for Inhalation, 80mg | Kamada-AAT for Inhalation, 160mg | Placebo
Number analyzed (Participants) | 11 | 11 | 11
nM | 113.17 [56.3 to 158.1] | 90.73 [37.3 to 369.7] | -4.02 [-9.8 to 4.9]
Statistical Analysis 1: Comparison: Kamada-AAT for Inhalation, 80mg vs Kamada-AAT for Inhalation, 160mg vs Placebo; Test type: Superiority; p < 0.0001, Kruskal-Wallis; p-value of Kruskal-Wallis test (3 groups: Kamada-AAT for Inhalation, 80mg,Kamada-AAT for Inhalation, 160mg and placebo)

4. Secondary Outcome: Change From Baseline in AAT-neutrophil Elastase (NE) Complexes in ELF
Description: Patients underwent a BAL procedure at baseline and 12 weeks and the fluid was analyzed to calculate the change from baseline in the concentration of complexes between AAT and neutrophil elastase in the ELF
Time Frame: 12 weeks from initiation of study drug
Measure: Median (95% Confidence Interval); unit: nM
Arm/Group | Kamada-AAT for Inhalation, 80mg | Kamada-AAT for Inhalation, 160mg | Placebo
Number analyzed (Participants) | 12 | 10 | 10
nM | 38.71 [8.4 to 66.8] | 46.225 [17.6 to 436.3] | 0 [-2 to 1.3]
Statistical Analysis 1: Comparison: Kamada-AAT for Inhalation, 80mg vs Kamada-AAT for Inhalation, 160mg; Test type: Superiority; p < 0.0001, Kruskal-Wallis; p-value of Kruskal-Wallis test (3 groups: Kamada-AAT for Inhalation, 80mg, Kamada-AAT for Inhalation, 160mg and placebo)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Kamada-AAT for Inhalation, 80mg | Kamada-AAT for Inhalation, 160mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 1/12 | 0/12
Other Adverse Events (participants affected / at risk) | 10/12 | 8/12 | 7/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Kamada-AAT for Inhalation, 80mg (N=12) | Kamada-AAT for Inhalation, 160mg (N=12) | Placebo (N=12)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — Community acquired pneumonia
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Kamada-AAT for Inhalation, 80mg (N=12) | Kamada-AAT for Inhalation, 160mg (N=12) | Placebo (N=12)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Lip swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0) | 1 (1)
Feeling jittery (General disorders) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 2 (2) | 2 (3)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Viral respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Pulmonary function test decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Urine analysis (Investigations) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (3) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (1) | 3 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal discharge discolouration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes